CLINICAL TRIAL: NCT00600886
Title: A Multicenter, Randomized, Blinded Study to Assess Safety and Efficacy of Pasireotide LAR vs. Octreotide LAR in Patients With Active Acromegaly
Brief Title: Safety and Efficacy of Pasireotide Long Acting Release (LAR) vs. Octreotide LAR in Patients With Active Acromegaly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSOM230C2305; 2007-001972-36 (EudraCT Number)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2015-01-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Acromegaly
Keywords: Acromegaly,; adult,; growth hormone,; insulin-like growth factor I,; somatostatin analogue
MeSH Terms: conditions — Acromegaly | interventions — pasireotide; Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pasireotide LAR (Experimental): Patients in this arm received Pasireotide LAR 40 mg im depot injection, blinded, once every 28 days (± 2 days) for 12 months. Dose could be down- or up-titrated to 20 or 60 mg, respectively. Patients who responded to Pasireotide LAR (i.e. the randomized treatment) at the end of the core (Month 12), continued Pasireotide LAR treatment in the extension. Patients who did not respond to Pasireotide LAR at the end of the core (Month 12) were allowed to switch to receive Octreotide LAR in the extension.
  Interventions: Drug: Pasireotide
- Octreotide LAR (Active Comparator): Patients in this arm received Octreotide LAR 20 mg im depot injection, blinded, once every 28 days (± 2 days) for 12 months. Dose could be down- or up-titrated to 10 or 30 mg, respectively. Patients who responded to Octreotide LAR (i.e. the randomized treatment) at the end of the core (Month 12) continued Octreotide LAR treatment in the extension (up to 2 years of treatment). Patients who did not respond to Octreotide LAR at the end of the core (Month 12) were allowed to switch to receive Pasireotide LAR in the extension.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Pasireotide — Pasireotide LAR - intramuscular (i.m.) depot injection given once every 28 days.
  Other Names: SOM230
  Arms: Pasireotide LAR
Drug: Octreotide — Octreotide LAR - i.m. depot injection given once every 28 days.
  Arms: Octreotide LAR

SUMMARY:
The patients received either Pasireotide LAR or Octreotide LAR for one year of treatment.

The objective of this study was to compare the proportion of patients with a reduction of mean GH level to <2.5 µg/L and the normalization of IGF-1 to within normal limits (age and sex related) between the two treatment groups (pasireotide LAR and octreotide LAR) at 12 months.

Following one year of treatment patients could proceed into the study extension.

Patients who did not respond to the treatment they were randomized to (based on month 12 assessment results) were switched to the other treatment arm at month 13.

ELIGIBILITY:
Inclusion criteria:

* Patients with active acromegaly (based on elevated GH and IGF-1 levels)
* Patients who have undergone one or more pituitary surgeries, but have not been treated medically, or de-novo patients presenting a visible pituitary adenoma on MRI and who refuse pituitary surgery or for whom pituitary surgery is contraindicated
* Patients for whom written informed consent to participate in the study has been obtained prior to any study related activity

Exclusion criteria:

* Patients who are being or were treated with octreotide, lanreotide, dopamine agonists or GH antagonists with the exception of a single dose of short-acting octrotide or short-acting dopamine agonists. In case of a single dose of short-acting octrotide, the dose should not be used to predict the response to the octretide treatment. The single dose of short-acting octreotide or short-acting dopamine agonists should not be administered in the 3 days prior to randomization
* Patients with compression of the optic chiasm causing any visual field defect
* Patients who have received pituitary irradiation within the last ten years prior to visit 1
* Poorly controlled diabetic patients

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2008-02-11 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (88):
- United States (14):
  - Cedars Sinai Medical Center The Pituitary Center, Los Angeles, California
  - University of California at Los Angeles Division of Endocrinology, Los Angeles, California
  - Stanford University Medical Center Stanford Cancer Center (3), Stanford, California
  - University of Florida SC, Gainesville, Florida
  - Johns Hopkins University School of Medicine Dept.ofJohnsHopkinsUniv., Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center Deptof Endocrinology&Diabetes, Ann Arbor, Michigan
  - Columbia University Medical Center- New York Presbyterian Dept. of CU Collegeof Phys&Sur, New York, New York
  - Northport VA Medical Center CSOM230C2305, Northport, New York
  - Oregon Health & Sciences University DeptofOregonHealth&Sciences(3), Portland, Oregon
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center Danziger Research Bldg., Dallas, Texas
  - University of Texas/MD Anderson Cancer Center Regulatory -12, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Swedish Medical Center Dept.ofSeattle Neuroscience(2), Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (6):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (2):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Bogota, Cundinamarca, Colombia
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Copenhagen
- France (7):
  - Novartis Investigative Site, Bois-Guillaume
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Piraeus
- Novartis Investigative Site, Budapest, Hungary
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (7):
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Netherlands (2):
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Alicante, Valencia
- Sweden (3):
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Erzurum
- United Kingdom (4):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Bronstein MD, Fleseriu M, Neggers S, Colao A, Sheppard M, Gu F, Shen CC, Gadelha M, Farrall AJ, Hermosillo Resendiz K, Ruffin M, Chen Y, Freda P; Pasireotide C2305 Study Group. Switching patients with acromegaly from octreotide to pasireotide improves biochemical control: crossover extension to a randomized, double-blind, Phase III study. BMC Endocr Disord. 2016 Apr 2;16:16. doi: 10.1186/s12902-016-0096-8. PMID 27039081
- [Derived] Shanik MH, Cao PD, Ludlam WH. HISTORICAL RESPONSE RATES OF SOMATOSTATIN ANALOGUES IN THE TREATMENT OF ACROMEGALY: A SYSTEMATIC REVIEW. Endocr Pract. 2016 Mar;22(3):350-6. doi: 10.4158/EP15913.RA. Epub 2015 Oct 5. PMID 26437217
- [Derived] Sheppard M, Bronstein MD, Freda P, Serri O, De Marinis L, Naves L, Rozhinskaya L, Hermosillo Resendiz K, Ruffin M, Chen Y, Colao A. Pasireotide LAR maintains inhibition of GH and IGF-1 in patients with acromegaly for up to 25 months: results from the blinded extension phase of a randomized, double-blind, multicenter, Phase III study. Pituitary. 2015 Jun;18(3):385-94. doi: 10.1007/s11102-014-0585-6. PMID 25103549
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?trialID=660

RESULTS

PARTICIPANT FLOW:
Period: Core Phase - Full Analysis Set (FAS)
Arm/Group | Pasireotide LAR | Octreotide LAR
Started | 176 | 182
Did Not Enter Extension | 29 | 29
Entered Extension, Crossed Over | 38 | 81
Entered Ext Continued Same Treatment | 74 | 46
Completed | 141 (Completed = anyone who did not discontinue prior to month 12.) | 156 (Completed = anyone who did not discontinue prior to month 12.)
Not Completed | 35 | 26
Not completed — Adverse Event | 14 | 6
Not completed — Protocol Violation | 7 | 8
Not completed — Lack of Efficacy | 5 | 8
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Administrative Problems | 2 | 0
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1
Period: Extension - Same Treatment (FAS)
Arm/Group | Pasireotide LAR | Octreotide LAR
Started | 74 (Started = anyone who entered the extension and continued the same treatment of Pasireotide LAR) | 46 (Started = anyone who entered the extension and continued the same treatment of Octreotide LAR)
Completed Study at Month 26 | 0 (Pas. LAR pts in Ext. were not considered completers at M26 as treatment could continue after M26.) | 31 (Per protocol, pts who received Octreotide LAR in ext. phase were not followed in the study after M26)
Completed Study After Month 26 | 28 (Completed = Pts who transferred to a roll-over protocol or commercial supply of Pasireotide LAR) | 4 (Received treatment and completed after M26: Recorded as protocol deviation)
Discontinued After Month 26 | 23 | 1 (Received treatment and discontinued after M26: Recorded as protocol deviation)
Discontinued Between M12 and M26 | 23 | 10
Completed | 28 (Completed= completed after M26, switched to commercial pasireotide LAR or entered roll-over protocol) | 35 (Completed = completed the study)
Not Completed | 46 | 11
Not completed — Withdrawal by Subject | 16 | 2
Not completed — Lack of Efficacy | 3 | 3
Not completed — Administrative Problems | 9 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Abnormal Lab Value (s) | 4 | 0
Not completed — Death | 1 | 1
Not completed — Condition no longer requires study drug | 6 | 0
Period: Extension - After Crossover (CAS)
Arm/Group | Pasireotide LAR | Octreotide LAR
Started | 81 (Started = anyone who entered the extension and crossed over to Pasireotide LAR) | 38 (Started = anyone who entered the extension and crossed over to Octreotide LAR)
Completed Study at Month 26 | 0 (Pas. LAR pts in Ext. were not considered completers at M26 as treatment could continue after M26.) | 25 (Per protocol, Pts who received Octreotide LAR in Ext. phase were not followed in study after M26)
Completed After Month 26 | 19 (Completed = Pts who transferred to a roll-over protocol or commercial supply of Pasireotide LAR) | 0 (Per protocol, pts who received Octreotide LAR in ext. phase were not followed in study after M26)
Discontinued Between M12 and M26 | 31 | 13
Discontinued After M26 | 31 | 0 (Per protocol, Pts who received Octreotide LAR in Ext. phase were not followed in study after M26)
Completed | 19 (Completed after month 26: transferred to a roll-over protocol or commercial supply of Pas.LAR) | 25 (Completed the study)
Not Completed | 62 | 13
Not completed — Adverse Event | 19 | 1
Not completed — Withdrawal by Subject | 19 | 4
Not completed — Lack of Efficacy | 13 | 4
Not completed — Administrative Problems | 4 | 4
Not completed — Subject no longer requires study drug | 3 | 0
Not completed — Abnormal Lab Value (s) | 3 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All patients who were randomized into the study. Patients were analyzed according to the treatment they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR | Octreotide LAR | Total
Number analyzed (Participants) | 176 | 182 | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (12.37) | 45.6 (12.97) | 45.4 (12.67)
Age, Customized [Number; unit: Participants]
  <65 Years | 168 | 167 | 335
  >=65 years | 8 | 15 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 95 | 186
  Male | 85 | 87 | 172

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Reduction of Mean GH Level to <2.5 μg/L and the Normalization of IGF-1
Description: Percentage of participants with a reduction of mean GH levels to <2.5μg/L (based on a 5-point 2-hour profile) and normalization of sex- and age-adjusted IGF-1.
  Post surgery = patients with prior surgery but no previous medical treatment for acromegaly De novo = patients with de novo disease who refused pituitary surgery or for whom pituitary surgery was contraindicated.
Time Frame: 12 months
Population: Full Analysis Set: All patients (Pts) who were randomized into the study. Pts were analyzed according to the treatment they were assigned to at randomization. Missing mean GH and/or IGF-1 levels at M12 were imputed using data obtained at or after M6 by the last observation carried forward method; otherwise, Pts were considered as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Pasireotide LAR (Core): Includes data from the 12-month blinded core phase for patients randomized to receive Pasireotide LAR.
- Octreotide LAR (Core): Includes data from the 12-month blinded core phase for patients randomized to receive Octreotide LAR.
Arm/Group | Pasireotide LAR (Core) | Octreotide LAR (Core)
Number analyzed (Participants) | 176 | 182
Percentage of Participants
  Overall | 31.3 [24.5 to 38.7] | 19.2 [13.8 to 25.7]
  Post Surgery: number analyzed (Participants) | 71 | 78
  Post Surgery | 39.4 [28.0 to 51.7] | 21.8 [13.2 to 32.6]
  De novo: number analyzed (Participants) | 105 | 104
  De novo | 25.7 [17.7 to 35.2] | 17.3 [10.6 to 26.0]
Statistical Analysis 1: Comparison: Pasireotide LAR (Core) vs Octreotide LAR (Core); Overall - All patients; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel adjusting for randomization stratification factor; Odds Ratio (OR) = 1.942, 95% CI 2-sided [1.190 to 3.168]
Statistical Analysis 2: Comparison: Pasireotide LAR (Core) vs Octreotide LAR (Core); Post surgery - patients with prior surgery but no previous medical treatment for acromegaly; Test type: Superiority or Other; Odds Ratio (OR) = 2.337, 95% CI 2-sided [1.140 to 4.790]
Statistical Analysis 3: Comparison: Pasireotide LAR (Core) vs Octreotide LAR (Core); De novo - patients with de novo disease who refused pituitary surgery or for whom pituitary surgery was contraindicated; Test type: Superiority or Other; Odds Ratio (OR) = 1.654, 95% CI 2-sided [0.846 to 3.234]

2. Secondary Outcome: Percentage of Participants With a Reduction of Mean GH Level to < 2.5μg/L
Description: Percentage of participants with a reduction of mean GH levels to < 2.5μg/L (based on a 5-point 2-hour profile).
  Post surgery = patients with prior surgery but no previous medical treatment for acromegaly De novo = patients with de novo disease who refused pituitary surgery or for whom pituitary surgery was contraindicated.
Time Frame: 12 Months
Population: FAS: All patients (Pts) who were randomized into the study. Pts were analyzed according to the treatment they were assigned to at randomization. Missing mean GH levels at Month 12 were imputed using data obtained at or after Month 6 by the LOCF (last observation carried forward) method; otherwise, Pts were considered as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR (Core) | Octreotide LAR (Core)
Number analyzed (Participants) | 176 | 182
Percentage of participants
  Overall | 48.3 [40.7 to 55.9] | 51.6 [44.1 to 59.1]
  Post surgery: number analyzed (Participants) | 71 | 78
  Post surgery | 52.1 [39.9 to 64.1] | 51.3 [39.7 to 62.8]
  De novo: number analyzed (Participants) | 105 | 104
  De novo | 45.7 [36.0 to 55.7] | 51.9 [41.9 to 61.8]

3. Secondary Outcome: Change From Baseline in Tumor Volume at 12 Months
Description: Absolute and percentage change from baseline in tumor volume (assessed by pituitary MRI) Post surgery = patients with prior surgery but no previous medical treatment for acromegaly De novo = patients with de novo disease who refused pituitary surgery or for whom pituitary surgery was contraindicated.
Time Frame: Baseline, 12 Months
Population: Full Analysis Set (FAS): All patients who were randomized into the study. Patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Pasireotide LAR (Core) | Octreotide LAR (Core)
Number analyzed (Participants) | 176 | 182
mm^3
  Overall at baseline: number analyzed (Participants) | 166 | 169
  Overall at baseline | 2420.7 (4159.21) | 2259.2 (3390.20)
  Overall % change at month 12: number analyzed (Participants) | 120 | 124
  Overall % change at month 12 | -39.7 (21.83) | -38.0 (24.47)
  Post surgery at baseline: number analyzed (Participants) | 70 | 74
  Post surgery at baseline | 2185.2 (2861.09) | 2196.5 (3922.08)
  Post surgery % change at month 12: number analyzed (Participants) | 44 | 52
  Post surgery % change at month 12 | -39.5 (20.60) | -39.0 (23.81)
  De novo at baseline: number analyzed (Participants) | 96 | 95
  De novo at baseline | 2592.4 (4901.99) | 2308.1 (2930.84)
  De novo % change at month 12: number analyzed (Participants) | 76 | 72
  De novo % change at month 12 | -39.9 (22.65) | -37.2 (25.07)
  Overall absolute change at month 12: number analyzed (Participants) | 121 | 128
  Overall absolute change at month 12 | -987.1 (2448.14) | -801.2 (1676.62)
  Post surgery abs. change at month 12: number analyzed (Participants) | 44 | 55
  Post surgery abs. change at month 12 | -873.7 (1282.06) | -713.8 (1708.20)
  De novo absolute change at month 12: number analyzed (Participants) | 77 | 73
  De novo absolute change at month 12 | -1051.9 (2919.18) | -867.1 (1661.24)

4. Secondary Outcome: Percentage of Participants With Normalization of IGF-1
Description: Percentage of participants with normalization of sex- and age-adjusted IGF-1. Post surgery = patients with prior surgery but no previous medical treatment for acromegaly De novo = patients with de novo disease who refused pituitary surgery or for whom pituitary surgery was contraindicated.
Time Frame: 12 Months
Population: Full Analysis Set: All patients (Pts) who were randomized into the study. Pts were analyzed according to the treatment they were assigned to at randomization. Missing IGF-1 levels at Month 12 were imputed using data obtained at or after Month 6 by the LOCF (last observation carried forward) method; otherwise, Pts were considered as nonresponders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR (Core) | Octreotide LAR (Core)
Number analyzed (Participants) | 176 | 182
Percentage of participants
  Overall | 38.6 [31.4 to 46.3] | 23.6 [17.7 to 30.5]
  Post surgery: number analyzed (Participants) | 71 | 78
  Post surgery | 50.7 [38.6 to 62.8] | 26.9 [17.5 to 38.2]
  De novo: number analyzed (Participants) | 105 | 104
  De novo | 30.5 [21.9 to 40.2] | 21.2 [13.8 to 30.3]

5. Secondary Outcome: Percentage of Participants With a Reduction of Mean GH Level to < 2.5μg/L and Normalization of IGF-1
Description: Percentage of participants with a reduction of mean GH levels to < 2.5μg/L (based on a 5-point 2-hour profile) and normalization of sex- and age-adjusted IGF-1.
  Denominator for time points up to Month 12 is the Full Analysis Set (FAS). Denominator for time points after Month 12 excludes patients who completed the core and did not enter the extension. Patients who discontinued were considered non-responders for the time points after discontinuation, patients who crossed over were considered non-responders for all time points after crossover. Analysis was based on data up to crossover (i.e., included data from both blinded core & ext. phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included.)
Time Frame: Months 3, 6, 9, 12, 16, 19, 22, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR (Core & Extension): Includes data from both blinded core and extension phase (up to Month 26) for patients who continued the same treatment (Pasireotide LAR) as in the core. For patients who switched from blinded Pasireotide LAR to Octreotide LAR treatment in the extension, only data collected before crossover is included.
- Octreotide LAR (Core & Extension): Includes data from both blinded core and extension phase (up to Month 26) for patients who continued the same treatment (Octreotide LAR) as in the core. For patients who switched from blinded Octreotide LAR to Pasireotide LAR treatment in the extension, only data collected before crossover is included.
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Percentage of participants
  Month 3 | 30.1 [23.4 to 37.5] | 21.4 [15.7 to 28.1]
  Month 6 | 30.1 [23.4 to 37.5] | 19.8 [14.3 to 26.3]
  Month 9 | 27.8 [21.4 to 35.1] | 23.1 [17.2 to 29.9]
  Month 12 | 29.0 [22.4 to 36.3] | 17.6 [12.3 to 23.9]
  Month 16: number analyzed (Participants) | 147 | 153
  Month 16 | 25.2 [18.4 to 33.0] | 12.4 [7.6 to 18.7]
  Month 19: number analyzed (Participants) | 147 | 153
  Month 19 | 23.1 [16.6 to 30.8] | 13.7 [8.7 to 20.2]
  Month 22: number analyzed (Participants) | 147 | 153
  Month 22 | 25.2 [18.4 to 33.0] | 16.3 [10.9 to 23.2]
  Month 25: number analyzed (Participants) | 147 | 153
  Month 25 | 24.5 [17.8 to 32.3] | 13.7 [8.7 to 20.2]

6. Secondary Outcome: Summary of Mean GH Values
Description: Mean GH levels (based on a 5-point profile over 2 hours). Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, Months 3, 6, 9, 12, 16, 19, 22, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
μg/L
  Baseline: number analyzed (Participants) | 167 | 178
  Baseline | 21.9 (32.14) | 18.8 (25.95)
  Month 3: number analyzed (Participants) | 164 | 173
  Month 3 | 6.3 (12.54) | 5.8 (12.87)
  Month 6: number analyzed (Participants) | 151 | 165
  Month 6 | 5.6 (11.47) | 5.2 (10.99)
  Month 9: number analyzed (Participants) | 136 | 157
  Month 9 | 4.9 (9.62) | 4.3 (9.70)
  Month 12: number analyzed (Participants) | 136 | 151
  Month 12 | 4.6 (9.51) | 4.5 (11.34)
  Month 16: number analyzed (Participants) | 64 | 38
  Month 16 | 2.3 (5.64) | 1.4 (1.49)
  Month 19: number analyzed (Participants) | 62 | 38
  Month 19 | 2.1 (5.68) | 1.5 (1.68)
  Month 22: number analyzed (Participants) | 60 | 39
  Month 22 | 2.1 (6.15) | 1.4 (1.43)
  Month 25: number analyzed (Participants) | 62 | 40
  Month 25 | 2.0 (5.02) | 1.2 (1.11)

7. Secondary Outcome: Time to First Response for Patients Achieving a Reduction of Mean GH Level to < 2.5 μg/L and Normalization of IGF-1 (No. of Responders: Pasireotite LAR = 81, Octreotide LAR = 63) )
Description: Time to first response for patients achieving a reduction of mean GH level to < 2.5 μg/L and normalization of IGF-1. Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Up to 26 months
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Weeks | 12.6 [12.3 to 13.0] | 12.4 [12.3 to 13.7]

8. Secondary Outcome: Severity Scores of Acromegaly Symptoms
Description: Severity scores of acromegaly symptoms (Headache, Fatigue, Perspiration, Paresthesias, Osteoarthralgia). Symptoms were scored from 0 (no symptom) to 4 (very severe). Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, Months 12, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
scores on a scale
  Headache - Baseline: number analyzed (Participants) | 175 | 181
  Headache - Baseline | 0.9 (1.05) | 1.0 (1.14)
  Fatigue - Baseline: number analyzed (Participants) | 175 | 181
  Fatigue - Baseline | 1.2 (1.13) | 1.4 (1.23)
  Perspiration - Baseline: number analyzed (Participants) | 175 | 181
  Perspiration - Baseline | 1.1 (1.21) | 1.3 (1.31)
  Paresthesia - Baseline: number analyzed (Participants) | 175 | 180
  Paresthesia - Baseline | 0.7 (1.00) | 0.8 (1.15)
  Osteoarthraliga - Baseline: number analyzed (Participants) | 174 | 178
  Osteoarthraliga - Baseline | 1.0 (1.05) | 1.3 (1.26)
  Headache - M12: number analyzed (Participants) | 138 | 149
  Headache - M12 | 0.5 (0.77) | 0.6 (0.79)
  Fatigue - M12: number analyzed (Participants) | 138 | 149
  Fatigue - M12 | 0.8 (0.95) | 0.7 (0.99)
  Perspiration - M12: number analyzed (Participants) | 138 | 149
  Perspiration - M12 | 0.4 (0.81) | 0.5 (0.91)
  Paresthesia - M12: number analyzed (Participants) | 138 | 149
  Paresthesia - M12 | 0.3 (0.63) | 0.4 (0.72)
  Osteoarthraliga - M12: number analyzed (Participants) | 137 | 149
  Osteoarthraliga - M12 | 0.5 (0.80) | 0.7 (1.00)
  Headache - M25: number analyzed (Participants) | 64 | 40
  Headache - M25 | 0.4 (0.61) | 0.6 (0.77)
  Fatigue - M25: number analyzed (Participants) | 64 | 40
  Fatigue - M25 | 0.5 (0.71) | 0.7 (0.89)
  Perspiration - M25: number analyzed (Participants) | 64 | 40
  Perspiration - M25 | 0.4 (0.72) | 0.4 (0.67)
  Paresthesia - M25: number analyzed (Participants) | 64 | 40
  Paresthesia - M25 | 0.2 (0.49) | 0.4 (0.67)
  Osteoarthraliga - M25: number analyzed (Participants) | 64 | 40
  Osteoarthraliga - M25 | 0.4 (0.79) | 0.8 (1.07)

9. Secondary Outcome: Ring Size
Description: Ring size (based on jeweler's finger gauge). Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, Months 12, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: ring zize
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
ring zize
  Baseline left hand (LH) 4th digit: number analyzed (Participants) | 112 | 115
  Baseline left hand (LH) 4th digit | 11.6 (2.00) | 11.8 (1.97)
  Baseline left hand 5th digit: number analyzed (Participants) | 21 | 18
  Baseline left hand 5th digit | 11.7 (2.82) | 12.4 (2.88)
  Baseline right hand (RH) 4th digit: number analyzed (Participants) | 23 | 29
  Baseline right hand (RH) 4th digit | 12.5 (2.01) | 11.4 (2.54)
  Baseline right hand 5th digit: number analyzed (Participants) | 5 | 8
  Baseline right hand 5th digit | 11.2 (3.35) | 11.3 (2.95)
  M12 LH 4th digit: number analyzed (Participants) | 97 | 102
  M12 LH 4th digit | 10.6 (2.05) | 11.1 (1.95)
  M12 LH 5th digit: number analyzed (Participants) | 12 | 10
  M12 LH 5th digit | 11.8 (1.81) | 12.4 (1.78)
  M12 RH 4th digit: number analyzed (Participants) | 21 | 25
  M12 RH 4th digit | 12.2 (2.12) | 11.3 (2.18)
  M12 RH 5th digit: number analyzed (Participants) | 5 | 6
  M12 RH 5th digit | 10.7 (3.96) | 10.5 (2.14)
  M25 LH 4th digit: number analyzed (Participants) | 49 | 33
  M25 LH 4th digit | 10.1 (2.12) | 11.1 (1.95)
  M25 LH 5th digit: number analyzed (Participants) | 5 | 2
  M25 LH 5th digit | 10.0 (2.45) | 14.3 (0.35)
  M25 RH 4th digit: number analyzed (Participants) | 8 | 4
  M25 RH 4th digit | 11.8 (1.98) | 10.9 (1.65)
  M25 RH 5th digit: number analyzed (Participants) | 2 | 1
  M25 RH 5th digit | 7.8 (4.60) | 7.5 (NA) — N/A = Not applicable for Std. Dev.

10. Secondary Outcome: Health-related Quality-of-life as Measured by the AcroQoL Questionnaire
Description: Acromegalyy quality of life (AcroQoL) total scores. The AcroQoL questionnaire is unidimensional and contains 22 items divided in two scales: one that evaluates physical aspects (eight items) and another one that evaluates psychological aspects (14 items). The scoring of the questionnaire was performed as specified by the instrument developers. Total scores range from 0 to 100. Higher scores represent better quality of life. Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, Months 12, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Score on a scale
  Baseline: number analyzed (Participants) | 173 | 178
  Baseline | 58.4 (19.97) | 55.6 (19.79)
  M12: number analyzed (Participants) | 136 | 148
  M12 | 65.7 (21.64) | 61.6 (21.01)
  M25: number analyzed (Participants) | 58 | 38
  M25 | 69.3 (18.76) | 62.9 (18.86)

11. Secondary Outcome: Summary of Prolactin Levels
Description: Prolactin Levels. Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, Months 12, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
μg/L
  Baseline | 20.6 (53.00) | 15.8 (22.05)
  M12: number analyzed (Participants) | 135 | 146
  M12 | 8.9 (19.24) | 11.7 (19.09)
  M25: number analyzed (Participants) | 63 | 40
  M25 | 5.4 (4.37) | 6.7 (4.63)

12. Secondary Outcome: Duration of Response for Patients Achieving a Reduction of Mean GH Level to <2.5 μg/L and the Normalization of IGF-1 at Month 12 (No. of Responders: Pasireotide LAR = 51, Octreotide LAR = 32)
Description: The duration of response is defined as the time from the date that patient first met and maintained the response criteria based on primary efficacy variable to the date that patient lost response status.
  Median and corresponding 95% CI are derived based on Kaplan-Meier method. Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Up to 26 months
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Weeks | 64.4 [52.1 to 100.4] | 64.6 [40.0 to 92.0]

13. Secondary Outcome: Pasireotide Trough Concentrations by Incident Dose
Description: Pasireotide LAR trough concentrations by incident dose (last dose administered prior to PK sample collection). PK observations with missing concentrations, missing dose, missing elapsed time or an elapsed time from previous injection outside of 28±2 days window were excluded.
  5 patients with evaluable PK data in the pasireotide arm received erroneously 20 mg pasireotide LAR at baseline.
Time Frame: Months 1 - 12
Population: PK analysis set: All patients with at least one LAR injection and one post-dose trough concentration data in core phase (up to month 12). No participants took the 60 mg dose in Months 1, 2 and 3, hence no data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Pasireotide LAR 20 mg: Patients in this arm received Pasireotide LAR 20 mg injection prior to PK sample collection.
- Pasireotide LAR 40 mg: Patients in this arm received Pasireotide LAR 40 mg injection prior to PK sample collection.
- Pasireotide LAR 60mg: Patients in this arm received Pasireotide LAR 60 mg injection prior to PK sample collection.
Arm/Group | Pasireotide LAR 20 mg | Pasireotide LAR 40 mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 172 | 172 | 172
ng/mL
  M1: number analyzed (Participants) | 5 | 146 | 0
  M1 | 4.65 (0.645) | 6.65 (3.641) |
  M2: number analyzed (Participants) | 6 | 135 | 0
  M2 | 2.88 (1.371) | 7.81 (3.505) |
  M3: number analyzed (Participants) | 2 | 135 | 0
  M3 | 3.39 (2.659) | 8.70 (5.402) |
  M4: number analyzed (Participants) | 3 | 88 | 49
  M4 | 3.93 (1.858) | 9.51 (5.487) | 13.48 (7.750)
  M5: number analyzed (Participants) | 4 | 77 | 56
  M5 | 5.22 (4.077) | 10.92 (6.017) | 13.42 (6.902)
  M6: number analyzed (Participants) | 3 | 71 | 57
  M6 | 2.87 (1.101) | 10.59 (6.216) | 13.08 (6.967)
  M7: number analyzed (Participants) | 3 | 69 | 60
  M7 | 2.29 (0.857) | 11.85 (7.781) | 14.76 (6.868)
  M8: number analyzed (Participants) | 3 | 63 | 70
  M8 | 3.65 (1.865) | 12.33 (7.619) | 15.88 (9.073)
  M9: number analyzed (Participants) | 4 | 59 | 65
  M9 | 4.80 (1.957) | 12.75 (8.604) | 16.03 (10.852)
  M10: number analyzed (Participants) | 5 | 61 | 59
  M10 | 5.66 (3.606) | 12.42 (7.252) | 16.01 (11.497)
  M11: number analyzed (Participants) | 5 | 53 | 65
  M11 | 5.10 (2.375) | 12.62 (6.920) | 16.31 (10.596)
  M12: number analyzed (Participants) | 4 | 45 | 58
  M12 | 4.54 (1.634) | 11.11 (6.489) | 16.16 (9.323)

14. Secondary Outcome: Octreotide Trough Concentrations by Incident Dose
Description: Octreotide LAR trough concentrations by incident dose (last dose administered prior to PK sample collection). PK observations with missing concentrations, missing dose, missing elapsed time or an elapsed time from previous injection outside of 28±2 days window were excluded.
Time Frame: Months 1 - 12
Population: PK analysis set: All patients with at least one LAR injection and one post-dose trough concentration data in core phase (up to month 12). No participants took the 30 mg dose in Months 1, 2 and 3, hence no data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Octreotide LAR 10mg: Patients in this arm received Octreotide LAR 10 mg injection prior to PK sample collection.
- Octreotide LAR 20 mg: Patients in this arm received Octreotide LAR 20 mg injection prior to PK sample collection.
- Octreotide LAR 30 mg: Patients in this arm received Octreotide LAR 30 mg injection prior to PK sample collection.
Arm/Group | Octreotide LAR 10mg | Octreotide LAR 20 mg | Octreotide LAR 30 mg
Number analyzed (Participants) | 178 | 178 | 178
ng/mL
  M1: number analyzed (Participants) | 0 | 153 | 0
  M1 |  | 0.86 (0.493) |
  M2: number analyzed (Participants) | 2 | 139 | 0
  M2 | 0.61 (0.280) | 1.21 (0.663) |
  M3: number analyzed (Participants) | 2 | 134 | 0
  M3 | 0.62 (0.107) | 1.29 (0.654) |
  M4: number analyzed (Participants) | 1 | 79 | 64
  M4 | 0.19 (NA) — N/A = Insufficient number of participants to calculate standard deviation. | 1.45 (0.653) | 1.55 (0.658)
  M5: number analyzed (Participants) | 0 | 63 | 82
  M5 |  | 1.65 (0.876) | 2.14 (1.156)
  M6: number analyzed (Participants) | 2 | 62 | 88
  M6 | 1.33 (0.754) | 1.58 (0.811) | 2.12 (0.990)
  M7: number analyzed (Participants) | 1 | 61 | 82
  M7 | 0.70 (NA) — N/A = Insufficient number of participants to calculate standard deviation. | 1.46 (0.704) | 2.14 (1.009)
  M8: number analyzed (Participants) | 0 | 50 | 88
  M8 |  | 1.55 (0.727) | 2.16 (1.127)
  M9: number analyzed (Participants) | 0 | 47 | 93
  M9 |  | 1.74 (1.013) | 2.20 (0.992)
  M10: number analyzed (Participants) | 0 | 49 | 82
  M10 |  | 1.66 (0.995) | 2.50 (1.194)
  M11: number analyzed (Participants) | 0 | 43 | 87
  M11 |  | 1.74 (0.890) | 2.39 (1.103)
  M12: number analyzed (Participants) | 1 | 37 | 76
  M12 | 0.30 (NA) — N/A = Insufficient number of participants to calculate standard deviation. | 1.58 (0.695) | 2.55 (1.252)

15. Secondary Outcome: Percentage of Participants With a Reduction of Mean GH Level to < 2.5μg/L and Normalization of IGF-1 After Crossover
Description: Percentage of participants with a reduction of mean GH levels to < 2.5μg/L (based on a 5-point 2-hour profile) and normalization of sex- and age-adjusted IGF-1. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). Denominator for all time points is the Crossover Analysis Set (CAS).
Time Frame: Months 3, 6, 9, 12 after crossover
Population: Crossover Analysis Set (CAS): All patients whose first dose in the extension is different from the first dose in the core.
  Patients were analyzed according to the crossover treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Crossed Over to Pasireotide LAR (Extension): Includes data from the blinded extension phase (up to Month 26) collected after the crossover time point for patients who crossed over from Octreotide LAR treatment in the core to Pasireotide LAR treatment in the extension phase.
- Crossed Over to Octreotide LAR (Extension): Includes data from the blinded extension phase (up to Month 26) collected after the crossover time point for patients who crossed over from Pasireotide LAR treatment in the core to Octreotide LAR treatment in the extension phase.
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
Percentage of participants
  M3 after crossover | 17.3 [9.8 to 27.3] | 2.6 [0.1 to 13.8]
  M6 after crossover | 21.0 [12.7 to 31.5] | 2.6 [0.1 to 13.8]
  M9 after crossover | 22.2 [13.7 to 32.8] | 5.3 [0.6 to 17.7]
  M12 after crossover | 17.3 [9.8 to 27.3] | 0.0 [NA to NA] — N/A = For zero proportions, confidence intervals were not calculated

16. Secondary Outcome: Percentage of Participants With a Reduction of Mean GH Level to < 2.5μg/L
Description: Percentage of participants with a reduction of mean GH levels to < 2.5μg/L (based on a 5-point 2-hour profile).
  Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included). Denominator for time points up to Month 12 is the Full Analysis Set. Denominator for time points after Month 12 excludes patients who completed the core and did not enter the extension. Patients who discontinued were considered non-responders for the time points after discontinuation, patients who crossed over were considered non-responders for all time points after crossover.
Time Frame: Months 3, 6, 9, 12, 16, 19, 22, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Percentage of participants
  M3 | 49.4 [41.8 to 57.1] | 43.4 [36.1 to 50.9]
  M6 | 45.5 [37.9 to 53.1] | 47.8 [40.4 to 55.3]
  M9 | 42.6 [35.2 to 50.3] | 46.2 [38.8 to 53.7]
  M12 | 43.2 [35.8 to 50.8] | 47.3 [39.8 to 54.8]
  M16: number analyzed (Participants) | 147 | 153
  M16 | 33.3 [25.8 to 41.6] | 22.2 [15.9 to 29.6]
  M19: number analyzed (Participants) | 147 | 153
  M19 | 36.7 [28.9 to 45.1] | 21.6 [15.3 to 28.9]
  M22: number analyzed (Participants) | 147 | 153
  M22 | 35.4 [27.7 to 43.7] | 22.2 [15.9 to 29.6]
  M25: number analyzed (Participants) | 147 | 153
  M25 | 35.4 [27.7 to 43.7] | 24.2 [17.6 to 31.8]

17. Secondary Outcome: Percentage of Participants With Normalization of IGF-1
Description: Percentage of participants with normalization of sex- and age-adjusted IGF-1. Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included). Denominator for time points up to Month 12 is the FAS. Denominator for time points after Month 12 excludes patients who completed the core and did not enter the extension. Patients who discontinued were considered non-responders for the time points after discontinuation, patients who crossed over were considered non-responders for all time points after crossover.
Time Frame: Months 3, 6, 9, 12, 16, 19, 22, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
Percentage of participants
  M3 | 35.2 [28.2 to 42.8] | 25.3 [19.1 to 32.2]
  M6 | 35.8 [28.7 to 43.4] | 24.2 [18.1 to 31.1]
  M9 | 34.1 [27.1 to 41.6] | 28.0 [21.6 to 35.1]
  M12 | 35.8 [28.7 to 43.4] | 22.0 [16.2 to 28.7]
  M16: number analyzed (Participants) | 147 | 153
  M16 | 29.9 [22.7 to 38.0] | 13.7 [8.7 to 20.2]
  M19: number analyzed (Participants) | 147 | 153
  M19 | 25.2 [18.4 to 33.0] | 15.7 [10.3 to 22.4]
  M22: number analyzed (Participants) | 147 | 153
  M22 | 25.9 [19.0 to 33.7] | 17.0 [11.4 to 23.9]
  M25: number analyzed (Participants) | 147 | 153
  M25 | 25.9 [19.0 to 33.7] | 14.4 [9.2 to 21.0]

18. Secondary Outcome: Change From Baseline in Tumor Volume
Description: Percentage change from baseline in tumor volume (assessed by pituitary MRI). Analysis was based on data up to crossover (i.e., included data from both blinded core and extension phase up to 26 Months for patients who continued the same treatment in the extension. For patients who switched to the other treatment, only data collected before crossover was included).
Time Frame: Baseline, months 6, 12, 19, 25
Population: Full Analysis Set: All patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Pasireotide LAR (Core & Extension) | Octreotide LAR (Core & Extension)
Number analyzed (Participants) | 176 | 182
mm^3
  Baseline: number analyzed (Participants) | 166 | 169
  Baseline | 2420.7 (4159.21) | 2259.2 (3390.20)
  M6: number analyzed (Participants) | 148 | 160
  M6 | 1614.1 (2536.46) | 1565.4 (2245.99)
  M12: number analyzed (Participants) | 125 | 138
  M12 | 1482.4 (2387.88) | 1390.4 (2179.93)
  M19: number analyzed (Participants) | 59 | 37
  M19 | 956.6 (1806.72) | 1009.9 (1578.75)
  M25: number analyzed (Participants) | 59 | 36
  M25 | 840.4 (1706.07) | 814.1 (1306.58)
  % change at M6: number analyzed (Participants) | 142 | 145
  % change at M6 | -29.9 (21.73) | -28.8 (20.22)
  % change at M12: number analyzed (Participants) | 120 | 124
  % change at M12 | -39.7 (21.83) | -38.0 (24.47)
  % change at M19: number analyzed (Participants) | 56 | 35
  % change at M19 | -48.9 (22.81) | -47.2 (24.08)
  % change at M25: number analyzed (Participants) | 54 | 34
  % change at M25 | -51.8 (20.81) | -55.0 (21.27)

19. Secondary Outcome: Percentage of Participants With a Reduction of Mean GH Level to < 2.5μg/L After Crossover
Description: Percentage of participants with a reduction of mean GH levels to < 2.5μg/L (based on a 5-point 2-hour profile). Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). Denominator for all time points is the Crossover Analysis Set (CAS).
Time Frame: Months 3, 6, 9, 12 after crossover
Population: CAS: All patients whose first dose in the extension is different from the first dose in the core. Patients were analyzed according to the crossover treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
Percentage of participants
  M3 after crossover | 49.4 [38.1 to 60.7] | 28.9 [15.4 to 45.9]
  M6 after crossover | 43.2 [32.2 to 54.7] | 31.6 [17.5 to 48.7]
  M9 after crossover | 54.3 [42.9 to 65.4] | 31.6 [17.5 to 48.7]
  M12 after crossover | 44.4 [33.4 to 55.9] | 23.7 [11.4 to 40.2]

20. Secondary Outcome: Percentage of Participants With Normalization of IGF-1 After Crossover
Description: Percentage of participants with normalization of sex- and age-adjusted IGF-1. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). Denominator for all time points is the Crossover Analysis Set (CAS).
Time Frame: Months 3, 6, 9, 12 after crossover
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
Percentage of participants
  M3 after crossover | 19.8 [11.7 to 30.1] | 7.9 [1.7 to 21.4]
  M6 after crossover | 30.9 [21.1 to 42.1] | 7.9 [1.7 to 21.4]
  M9 after crossover | 29.6 [20.0 to 40.8] | 10.5 [2.9 to 24.8]
  M12 after crossover | 27.2 [17.9 to 38.2] | 5.3 [0.6 to 17.7]

21. Secondary Outcome: Summary of Mean GH Values After Crossover
Description: Mean GH levels (based on a 5-point profile over 2 hours). Extension baseline was defined as last measurement prior to the start of crossover treatment. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over).
Time Frame: Extension baseline, months 3, 6, 9, 12 after crossover
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
μg/L
  Ext. Baseline: number analyzed (Participants) | 78 | 33
  Ext. Baseline | 5.9 (15.02) | 7.1 (9.80)
  M3 after crossover: number analyzed (Participants) | 72 | 36
  M3 after crossover | 5.9 (19.70) | 9.8 (17.09)
  M6 after crossover: number analyzed (Participants) | 68 | 32
  M6 after crossover | 4.8 (14.51) | 9.8 (20.49)
  M9 after crossover: number analyzed (Participants) | 61 | 32
  M9 after crossover | 2.6 (3.03) | 8.7 (19.26)
  M12 after crossover: number analyzed (Participants) | 57 | 29
  M12 after crossover | 2.5 (2.47) | 10.4 (26.00)

22. Secondary Outcome: Change From Extension Baseline in Tumor Volume After Crossover
Description: Percentage change from extension baseline in tumor volume (assessed by pituitary MRI).
  Extension baseline was defined as last assessment prior to the administration of the new treatment after crossover. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over).
Time Frame: Extension baseline, months 6, 12 after crossover
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
mm^3
  Ext. Baseline: number analyzed (Participants) | 73 | 32
  Ext. Baseline | 1420.9 (1914.58) | 1809.6 (2579.25)
  Value at M6 after crossover: number analyzed (Participants) | 65 | 31
  Value at M6 after crossover | 1027.5 (1282.42) | 1794.9 (2823.08)
  % change - M6 after crossover: number analyzed (Participants) | 59 | 27
  % change - M6 after crossover | -18.1 (17.68) | -12.3 (24.11)
  Value at M12 after crossover: number analyzed (Participants) | 51 | 30
  Value at M12 after crossover | 949.0 (1169.49) | 1610.4 (2666.66)
  % change - M12 after crossover: number analyzed (Participants) | 46 | 26
  % change - M12 after crossover | -24.7 (25.20) | -17.9 (27.80)

23. Secondary Outcome: Severity Scores of Acromegaly Symptoms After Crossover
Description: Severity scores of acromegaly symptoms (Headache, Fatigue, Perspiration, Paresthesias, Osteoarthralgia).
  Symptoms were scored from 0 (no symptom) to 4 (very severe). Extension baseline was defined as last measurement prior to the start of crossover treatment. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over).
Time Frame: Extension baseline, month 12 after crossover
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
scores on a scale
  Headache: Ext. BL | 0.6 (0.89) | 0.4 (0.60)
  Headache: M12 after crossover: number analyzed (Participants) | 60 | 32
  Headache: M12 after crossover | 0.5 (0.83) | 0.7 (0.79)
  Fatigue: Ext. BL | 0.8 (1.07) | 0.7 (0.76)
  Fatigue: M12 after crossover: number analyzed (Participants) | 60 | 32
  Fatigue: M12 after crossover | 0.8 (0.91) | 0.7 (0.68)
  Perspiration: Ext. BL | 0.5 (0.85) | 0.6 (0.86)
  Perspiration: M12 after crossover: number analyzed (Participants) | 60 | 32
  Perspiration: M12 after crossover | 0.6 (0.98) | 0.5 (0.80)
  Paresthesia: Ext. BL | 0.4 (0.75) | 0.4 (.054)
  Paresthesia: M12 after crossover: number analyzed (Participants) | 60 | 32
  Paresthesia: M12 after crossover | 0.3 (0.56) | 0.4 (0.76)
  Osteoarthralgia: Ext. BL | 0.6 (0.91) | 0.6 (0.79)
  Osteoarthralgia: M12 after crossover: number analyzed (Participants) | 60 | 32
  Osteoarthralgia: M12 after crossover | 0.5 (0.89) | 0.7 (0.86)

24. Secondary Outcome: Ring Size After Crossover
Description: Ring size (based on jeweler's finger gauge). Extension baseline was defined as last measurement prior to the start of crossover treatment. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). BL = baseline, LH = left hand, RH = right hand, CO = crossover
Time Frame: Extension baseline, month 12 after crossover
Population: CAS: All patients whose first dose in the extension is different from the first dose in the core. Patients were analyzed according to the crossover treatment received. In the extension baseline, no participant had ring size on their right hand measured at the 5th digit, hence no data.
Measure: Mean (Standard Deviation); unit: ring size
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
ring size
  Ext. BL LH 4th digit: number analyzed (Participants) | 55 | 26
  Ext. BL LH 4th digit | 11.2 (2.10) | 11.0 (1.87)
  Ext. BL LH 5th digit: number analyzed (Participants) | 6 | 5
  Ext. BL LH 5th digit | 11.6 (1.88) | 12.3 (2.46)
  Ext. BL RH 4th digit: number analyzed (Participants) | 15 | 7
  Ext. BL RH 4th digit | 11.4 (2.42) | 12.4 (2.11)
  Ext. BL RH 5th digit: number analyzed (Participants) | 3 | 0
  Ext. BL RH 5th digit | 10.7 (2.31) |
  M12 after CO LH 4th digit: number analyzed (Participants) | 42 | 24
  M12 after CO LH 4th digit | 10.9 (2.27) | 11.2 (2.01)
  M12 after CO LH 5th digit CO: number analyzed (Participants) | 4 | 4
  M12 after CO LH 5th digit CO | 11.9 (2.14) | 12.5 (1.35)
  M12 after CO RH 4th digit: number analyzed (Participants) | 11 | 4
  M12 after CO RH 4th digit | 11.6 (2.95) | 11.4 (2.56)
  M12 after CO RH 5th digit: number analyzed (Participants) | 2 | 0
  M12 after CO RH 5th digit | 11.5 (0.00) |

25. Secondary Outcome: Health-related Quality-of-life as Measured by the AcroQoL Questionnaire After Crossover
Description: AcroQoL total scores. The AcroQoL questionnaire is unidimensional and contains 22 items divided in two scales: one that evaluates physical aspects (eight items) and another one that evaluates psychological aspects (14 items). The scoring of the questionnaire was performed as specified by the instrument developers. Extension baseline was defined as last measurement prior to the start of crossover treatment. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). Total scores range from 0 to 100. Higher scores represent better quality of life.
Time Frame: Extension baseline, months 12 after crossover
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
scores on a scale
  Ext. Baseline: number analyzed (Participants) | 79 | 34
  Ext. Baseline | 58.9 (23.11) | 59.8 (22.40)
  M12 after crossover: number analyzed (Participants) | 57 | 30
  M12 after crossover | 60.3 (24.34) | 61.2 (21.62)

26. Secondary Outcome: Summary of Prolactin Levels After Crossover
Description: Prolactin (PRL) levels. Analysis was based on data after crossover (i.e., included data from blinded extension phase collected after the crossover time point for patients who crossed over). Extension baseline was defined as last measurement prior to the start of crossover treatment.
Time Frame: Extension baseline, month 12 after crossover
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Crossed Over to Pasireotide LAR (Extension) | Crossed Over to Octreotide LAR (Extension)
Number analyzed (Participants) | 81 | 38
μg/L
  Ext. Baseline: number analyzed (Participants) | 78 | 34
  Ext. Baseline | 11.9 (18.42) | 15.7 (36.76)
  M12 after crossover: number analyzed (Participants) | 60 | 31
  M12 after crossover | 7.5 (8.95) | 16.1 (25.37)

ADVERSE EVENTS:
Description: Safety Set (SS): all pts given drug with post baseline assessment. Pts analyzed as per treatment (trt) 1st received. 2 pts randomized to Oct. LAR who received Pas. LAR as 1st dose were included in Pas. grp.
  Crossover Analysis Set (CAS): all pts with 1st dose in Ext. different from 1st dose in Core. Pts were analyzed acc. to crossover trt received.
Groups:
- Pasireotide LAR - up to 26 Months: Includes data from both blinded core and extension phase (up to Month 26 cutoff date of 29-Dec-2011) for patients who continued the same treatment (Pasireotide LAR) as in the core. For patients who switched from blinded Pasireotide LAR to Octreotide LAR treatment, only data collected before crossover is included.
- Octreotide LAR - up to 26 Months: Includes data from both blinded core and extension phase (up to Month 26 cutoff date of 29-Dec-2011) for patients who continued the same treatment (Octreotide LAR) as in the core. For patients who switched from blinded Octreotide LAR to Pasireotide LAR treatment, only data collected before crossover is included.
- Crossed Over to Pasireotide LAR - up to 26 Months: Includes all data in the extension phase (up to 26-Month cutoff date of 29-Dec-2011) collected after the crossover time point for patients who crossed over from Octreotide LAR in the core to Pasireotide LAR treatment in the extension phase.
- Crossed Over to Octreotide LAR - up to 26 Months: Includes all data in the extension phase (up to 26-Month cutoff date of 29-Dec-2011) collected after the crossover time point for patients who crossed over from Pasireotide LAR in the core to Octreotide LAR treatment in the extension phase.
- Pasireotide LAR - up to EOS: Includes data from both core and extension phase (up to End-of-study date of 11-Mar-2016) for patients who continued the same treatment (Pasireotide LAR) as in the core. For patients who switched from blinded Pasireotide LAR to Octreotide LAR treatment, only data collected before crossover is included.
  Per protocol, patients on Pasireotide LAR could continue to receive open-label Pasireotide LAR after treatment unblinding at Month 26, whereas those on Octreotide LAR were not followed after Month 26.
- Crossed Over to Pasireotide LAR - up to EOS: Includes all data in the extension phase (up to End-of-study date of 11-Mar-2016) collected after the crossover time point for patients who crossed over from Octreotide LAR in the core to Pasireotide LAR treatment in the extension phase.
  Per protocol, patients on Pasireotide LAR could continue to receive open-label Pasireotide LAR after treatment unblinding at Month 26, whereas those on Octreotide LAR were not followed after Month 26.
Arm/Group | Pasireotide LAR - up to 26 Months | Octreotide LAR - up to 26 Months | Crossed Over to Pasireotide LAR - up to 26 Months | Crossed Over to Octreotide LAR - up to 26 Months | Pasireotide LAR - up to EOS | Crossed Over to Pasireotide LAR - up to EOS
Serious Adverse Events (participants affected / at risk) | 35/178 | 28/180 | 8/81 | 6/38 | 37/178 | 12/81
Other Adverse Events (participants affected / at risk) | 169/178 | 161/180 | 74/81 | 33/38 | 170/178 | 76/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR - up to 26 Months (N=178) | Octreotide LAR - up to 26 Months (N=180) | Crossed Over to Pasireotide LAR - up to 26 Months (N=81) | Crossed Over to Octreotide LAR - up to 26 Months (N=38) | Pasireotide LAR - up to EOS (N=178) | Crossed Over to Pasireotide LAR - up to EOS (N=81)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acromegaly (Endocrine disorders) | 2 | 0 | 0 | 0 | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toxic nodular goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Concomitant disease progression (General disorders) | 2 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 5 | 4 | 2 | 1 | 5 | 3
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 3 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Catatonia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR - up to 26 Months (N=178) | Octreotide LAR - up to 26 Months (N=180) | Crossed Over to Pasireotide LAR - up to 26 Months (N=81) | Crossed Over to Octreotide LAR - up to 26 Months (N=38) | Pasireotide LAR - up to EOS (N=178) | Crossed Over to Pasireotide LAR - up to EOS (N=81)
Anaemia (Blood and lymphatic system disorders) | 14 | 10 | 6 | 1 | 19 | 8
Sinus bradycardia (Cardiac disorders) | 13 | 10 | 2 | 1 | 15 | 3
Cataract (Eye disorders) | 0 | 1 | 1 | 2 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 8 | 1 | 0 | 0 | 10 | 0
Abdominal distension (Gastrointestinal disorders) | 21 | 22 | 0 | 2 | 21 | 0
Abdominal pain (Gastrointestinal disorders) | 33 | 43 | 3 | 1 | 36 | 4
Abdominal pain upper (Gastrointestinal disorders) | 12 | 17 | 3 | 0 | 14 | 4
Constipation (Gastrointestinal disorders) | 10 | 19 | 4 | 1 | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 70 | 79 | 20 | 6 | 72 | 26
Dyspepsia (Gastrointestinal disorders) | 8 | 7 | 3 | 1 | 9 | 4
Flatulence (Gastrointestinal disorders) | 10 | 11 | 0 | 0 | 11 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 2 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 27 | 41 | 8 | 2 | 29 | 10
Vomiting (Gastrointestinal disorders) | 19 | 15 | 3 | 1 | 22 | 4
Fatigue (General disorders) | 20 | 21 | 6 | 3 | 21 | 7
Injection site pain (General disorders) | 13 | 9 | 0 | 1 | 14 | 0
Pyrexia (General disorders) | 8 | 10 | 1 | 0 | 11 | 2
Biliary dilatation (Hepatobiliary disorders) | 5 | 8 | 4 | 1 | 5 | 5
Cholelithiasis (Hepatobiliary disorders) | 56 | 69 | 18 | 6 | 59 | 23
Gallbladder polyp (Hepatobiliary disorders) | 5 | 3 | 4 | 2 | 8 | 5
Hepatic steatosis (Hepatobiliary disorders) | 10 | 11 | 6 | 3 | 11 | 6
Bronchitis (Infections and infestations) | 10 | 4 | 0 | 0 | 13 | 2
Influenza (Infections and infestations) | 16 | 11 | 3 | 3 | 18 | 4
Nasopharyngitis (Infections and infestations) | 32 | 29 | 13 | 7 | 34 | 15
Sinusitis (Infections and infestations) | 6 | 6 | 2 | 1 | 9 | 3
Upper respiratory tract infection (Infections and infestations) | 16 | 7 | 3 | 2 | 20 | 5
Urinary tract infection (Infections and infestations) | 9 | 12 | 5 | 0 | 11 | 10
Alanine aminotransferase increased (Investigations) | 15 | 10 | 3 | 0 | 16 | 5
Aspartate aminotransferase increased (Investigations) | 12 | 8 | 3 | 0 | 13 | 5
Blood bilirubin increased (Investigations) | 9 | 5 | 1 | 1 | 11 | 3
Blood creatine phosphokinase increased (Investigations) | 25 | 24 | 7 | 6 | 27 | 8
Blood glucose increased (Investigations) | 17 | 6 | 8 | 0 | 18 | 8
Blood thyroid stimulating hormone decreased (Investigations) | 4 | 2 | 1 | 2 | 5 | 1
Blood triglycerides increased (Investigations) | 4 | 4 | 2 | 4 | 8 | 2
Blood uric acid increased (Investigations) | 6 | 3 | 1 | 0 | 10 | 2
Electrocardiogram QT prolonged (Investigations) | 9 | 10 | 3 | 0 | 10 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 11 | 1 | 0 | 3 | 2
Glycosylated haemoglobin increased (Investigations) | 11 | 5 | 7 | 0 | 12 | 9
Insulin-like growth factor decreased (Investigations) | 1 | 0 | 1 | 0 | 2 | 5
Lipase increased (Investigations) | 10 | 13 | 3 | 2 | 11 | 3
Weight decreased (Investigations) | 9 | 8 | 2 | 0 | 9 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 38 | 8 | 18 | 3 | 40 | 19
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 | 1 | 5 | 0 | 3 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 4 | 2 | 1 | 10 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 55 | 18 | 25 | 5 | 56 | 29
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 4 | 5 | 2 | 5 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 2 | 1 | 0 | 9 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 14 | 7 | 2 | 14 | 8
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 12 | 0 | 3 | 0 | 12 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 25 | 10 | 2 | 24 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 21 | 6 | 3 | 24 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 10 | 7 | 1 | 10 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 1 | 1 | 9 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 2 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 8 | 6 | 1 | 16 | 6
Dizziness (Nervous system disorders) | 21 | 20 | 7 | 4 | 22 | 9
Headache (Nervous system disorders) | 41 | 49 | 17 | 5 | 42 | 20
Paraesthesia (Nervous system disorders) | 8 | 4 | 0 | 1 | 9 | 0
Anxiety (Psychiatric disorders) | 9 | 7 | 1 | 0 | 11 | 2
Insomnia (Psychiatric disorders) | 8 | 9 | 2 | 1 | 12 | 4
Haematuria (Renal and urinary disorders) | 6 | 2 | 1 | 2 | 8 | 2
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 17 | 1 | 1 | 16 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 15 | 3 | 1 | 9 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 36 | 3 | 1 | 34 | 4
Hypertension (Vascular disorders) | 18 | 16 | 5 | 3 | 21 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.